CLINICAL TRIAL: NCT04419610
Title: Investigating the Relationship Between the Renin Angiotensin System and the Coagulopathy Associated With COVID-19
Brief Title: RAS and Coagulopathy in COVID19
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 283093
Record Dates: First submitted 2020-04-16; First posted 2020-06-05 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: COVID
MeSH Terms: interventions — Sar-Arg-Val-Tyr-Ile-His-Pro-Ala-OH; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with confirmed/suspected C19 given intervention (Experimental): Intravenous infusion of either placebo or TRV027 at 12mg/hr. Treatment will continue until discharge or for 7 days (whichever is sooner).
  Interventions: Biological: TRV027
- Patients with confirmed/suspected C19 given no intervention (Placebo Comparator): Saline infusion.
  Interventions: Other: sodium chloride 0.9%

INTERVENTIONS:
Biological: TRV027 — peptide for infusion
  Arms: Patients with confirmed/suspected C19 given intervention
Other: sodium chloride 0.9% — placebo comparator for infusion
  Arms: Patients with confirmed/suspected C19 given no intervention

SUMMARY:
To determine whether the coagulopathy associated with COVID-19 infection is driven by overactivation of the renin angiotensin system (RAS)

DETAILED DESCRIPTION:
The proposed study will be run as a double-blind, randomized controlled experimental medicine study in male and female hospitalised (n=60) aged 18 or over, with confirmed COVID-19 infection. Patients who are admitted due to confirmed COVID-19 infection will be screened with a routine medical assessment (see Table 1) and enrolled if they meet the eligibility criteria. Subjects will be block randomised based on age to continuous intravenous infusion of placebo or TRV027 for 7 days.

Day 1 procedures can occur on the same day of screening and include a venous blood test prior to commencing an intravenous infusion of either placebo or TRV027 at 12mg/hr. The infusions will continue for 7 days. Venous blood tests will be repeated at days 3, 5 and 8, amounting to approximately 120mLs of blood in total over the 8-day period.

Once the infusion has finished, the subjects will remain in hospital for a further 24 hours for vital signs and adverse event monitoring. If a subject exits the trial before the 7-day infusion finishes, they will be advised to remain in hospital for a 24 hour period for monitoring. Subjects will be followed up on Day 30 either via telephone or via medical records.

. The role of the renin angiotensin system (RAS) in COVID-19 infection has been widely discussed for two reasons. First, SARS-COV-2, the virus causing COVID-19, invades type II pneumocytes in the lung by binding to an enzyme called angiotensin converting enzyme 2 (ACE2). As the virus enters the cell, via one of its receptors, ACE2, it is thought that this is internalised and is hence unable to perform its physiological action of converting Angiotensin II (AngII) to Ang(1-7). Second, it has been noted that severe COVID-19 infection has many features which are strikingly similar to the effects of overactivation of the RAS. Indeed, these features are apparent in preclinical models using AngII infusions and include lung injury, lung inflammation, myocardial microinfarcts, characteristic glomerular thrombosis and coagulopathy. The coagulopathy is particularly noteworthy given an early increase in D-Dimer has very high positive predictor value for death in COVID-19, and D-dimer concentrations are unusually high in COVID-19, over and above what would be expected for an acute phase response or a pneumonia caused by a respiratory virus such as influenza.

AngII and Ang(1-7) affect various aspects of the coagulation system including platelets and endothelial cells, and we therefore hypothesise that overaction of RAS is partly responsible for the coagulopathy present in COVID-19 infection. Because the over activation of the RAS in COVID-19 infection is due to both Angiotensin II excess and Ang(1-7) depletion, standard tools to modulate RAS (angiotensin converting enzyme inhibitors and angiotensin receptor blockers) cannot be used to test this hypothesis as they address the Angiotensin II excess, but not the Ang(1-7) depletion. TRV027 is a similar peptide to Ang(1-7) but is a much more potent biased agonist at AT1R than Ang(1-7) and would be expected to oppose the effects of AngII accumulation, and functionally correct the Ang(1-7) deficiency. Hence it is an appropriate tool to examine the link between RAS activation and coagulopathy in the context of COVID-19 infection.

ELIGIBILITY:
INCLUSION CRITERIA

A subject will be eligible for inclusion in this study only if all of the following criteria apply at the time of screening:

1. Hospitalised with confirmed COVID-19 infection.
2. Screened within 96hrs of SARS-COV-2 positive PCR.
3. Age 18 or over
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
5. Systolic blood pressure between 100 and 180

EXCLUSION CRITERIA

A subject will not be eligible for inclusion in this study if any of the following criteria apply at the time of screening:

1. Any unrelated clinical condition, which, in the opinion of the investigator, may affect D-dimer during the course of the study, independent of COVID-19 infection, e.g. subsets of cancers and coagulopathies.
2. Concomitant medication which inhibit the action of TRV027 (ARB's).
3. Any clinically significant medical conditions that in the opinion of the investigator would compromise subjects' safety or compliance with study procedures.
4. Any clinical condition which in the opinion of the principal investigator would compromise the scientific integrity of the study
5. Unwillingness or inability to follow the procedures outlined in the protocol.
6. Subject is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DAVID OWEN, Principal Investigator — National Health Service, United Kingdom; Katrina Pollock, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robbins AJ, Che Bakri NA, Toke-Bjolgerud E, Edwards A, Vikraman A, Michalsky C, Fossler M, Lemm NM, Medhipour S, Budd W, Gravani A, Hurley L, Kapil V, Jackson A, Lonsdale D, Latham V, Laffan M, Chapman N, Cooper N, Szydlo R, Boyle J, Pollock KM, Owen D. The effect of TRV027 on coagulation in COVID-19: A pilot randomized, placebo-controlled trial. Br J Clin Pharmacol. 2023 Apr;89(4):1495-1501. doi: 10.1111/bcp.15618. Epub 2022 Dec 14. PMID 36437688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Started | 15 | 13
Completed | 10 | 11
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — discharged early | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Median (Full Range); unit: years] | 67 [47 to 89] | 70 [43 to 79] | 68.5 [43 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 5 | 2 | 7
  Mixed | 1 | 0 | 1
  Asian | 0 | 3 | 3
  Black | 0 | 2 | 2
  Other | 7 | 5 | 12
  Not reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Coagulopathy Associated With COVID-19
Description: Change from Day 1 (Baseline) in D-dimer Levels at Day 3
Time Frame: Day 1 (baseline) and Day 3).
Population: Incomplete analysis set
Measure: Median (Full Range); unit: ng/mL FEU
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
ng/mL FEU | -313 [-1253 to 822] | -129.5 [-365 to 710]

2. Secondary Outcome: Markers of Dysregulation of Coagulation System
Description: Change from Day 1 (Baseline) in platelet count Levels at Day 3 (10E9 platelets/L)
Time Frame: Day 1 (baseline) and Day 3
Measure: Median (Full Range); unit: 10E9 platelets/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
10E9 platelets/L | 25 [-12 to 129] | 28.5 [-113 to 107]

3. Secondary Outcome: Markers of Dysregulation of Coagulation System Change From Baseline
Description: Activated Partial Thromboplastin Time (aPTT) - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (Day 1) to Day 3
Measure: Median (Full Range); unit: SECONDS
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
SECONDS | -1.3 [-5.2 to 2.3] | -0.5 [-4.8 to 2.7]

4. Secondary Outcome: Markers of Dysregulation of Coagulation System
Description: INR - Change from Baseline (day 1) to Day 3:
  INR (International Normalised Ratio)
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: Unitless RATIO
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
Unitless RATIO | 1.25 [-1.6 to 3.6] | 0 [0 to 0.1]

5. Secondary Outcome: Markers of Dysregulation of Coagulation System
Description: fibrinogen (g/L) -Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: g/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
g/L | -0.67 [-2.8 to 1.68] | -0.94 [-1.81 to 2.11]

6. Secondary Outcome: Markers of Dysregulation of Coagulation System
Description: Ferritin Ug/mL -Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: ug/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
ug/L | 52.5 [-324 to 838] | -14 [-572 to 886]

7. Secondary Outcome: Markers of Dysregulation of RAS
Description: Plasma Renin activity (nmol/L/h) -Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: NMOL/L/h
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
NMOL/L/h | 0 [0 to 0] | -0.9 [-3.3 to 0.1]

8. Secondary Outcome: Markers of Haemolysis/Inflammation
Description: Total bilirubin (umol/L) -Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: UMOL/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
UMOL/L | -0.5 [-4 to 2] | 0 [-4 to 2]

9. Secondary Outcome: Markers of Haemolysis/Inflammation
Description: LDH u/L -Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: u/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
u/L | -17 [-217 to 270] | 1 [-151 to 102]

10. Secondary Outcome: Markers of Haemolysis/Inflammation
Description: Haptoglobin g/L - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: g/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
g/L | 0 [-1.09 to 0.08] | 0.13 [0 to 0.74]

11. Secondary Outcome: Markers of Inflammation (Bacterial Sepsis)
Description: Pro-calcitonin ug/L - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: ug/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
ug/L | 0 [-0.03 to 0.16] | 0 [-1.12 to 0.03]

12. Secondary Outcome: Markers of Organ Dysregulation - Kidney
Description: Creatinine (umol/L) - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: UMOL/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
UMOL/L | -4 [-16 to 11] | -5 [-14 to 10]

13. Secondary Outcome: Markers of Dysregulation of Cardiovascular System
Description: BNP (B-type natriuetic Peptide) ng/L - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: ng/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
ng/L | 60 [-5 to 762] | -19 [-66 to 62]

14. Secondary Outcome: Markers of Dysregulation of Cardiovascular System
Description: Troponin ng/L - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: ng/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
ng/L | -2.5 [-50 to 0] | -2.5 [-3 to 0]

15. Secondary Outcome: Marker of Dysregulation of Endocrine System
Description: glucose mmol/L - Change from Baseline (day 1) to Day 3
Time Frame: Baseline (day 1) to Day 3
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
Number analyzed (Participants) | 11 | 10
mmol/L | -1.1 [-2 to 0.1] | -0.00 [-4.7 to 3.8]

ADVERSE EVENTS:
Time Frame: Day 1 to day 7 and day 30 - 7 days of infused drug and follow up call on day 30
Arm/Group | Patients With Confirmed/Suspected C19 Given Intervention | Patients With Confirmed/Suspected C19 Given no Intervention
All-Cause Mortality (participants affected / at risk) | 2/15 | 1/13
Serious Adverse Events (participants affected / at risk) | 5/15 | 3/13
Other Adverse Events (participants affected / at risk) | 3/15 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Confirmed/Suspected C19 Given Intervention (N=15) | Patients With Confirmed/Suspected C19 Given no Intervention (N=13)
severe COVID 19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
confusion (Nervous system disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Confirmed/Suspected C19 Given Intervention (N=15) | Patients With Confirmed/Suspected C19 Given no Intervention (N=13)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
injection site reaction (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04419610/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04419610/SAP_003.pdf